CLINICAL TRIAL: NCT06517953
Title: A Phase II Study to Assess Befotertinib and Icotinib as First-Line Treatment in Patients With Locally Advanced or Metastatic NSCLC and Uncommon EGFR Mutation(IcomBine, GASTO-10114)
Brief Title: Befotertinib and Icotinib for NSCLC With Uncommon EGFR Mutations
Acronym: IcomBine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Hou, Principal Investigator, Sun Yet-Sen University Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2024-002
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer Metastatic; EGFR G719X; EGFR L861Q; EGFR S768I
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib + Befotertinib (Experimental): orally Icotinib 125mg Tid plus orally Befotertinib 100mg qd until progression disease
  Interventions: Drug: Icotinib; Drug: Befotertinib

INTERVENTIONS:
Drug: Icotinib — An orally first-generation EGFR inhibitior.
  Other Names: Conmana
Drug: Befotertinib — An orally available, irreversible, third-generation，mutant-selective epidermal growth factor receptor（EGFR）inhibitor. Befotertinib combine with icotinib means that both drugs will be given together until disease progression or meet the discontinuation criteria.
  Other Names: D-0316

SUMMARY:
This research study aims to explore the combination of two targeted drugs as first-line treatment for Non-Small Cell Lung Cancer (NSCLC) with uncommon EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Pathologically confirmed adenocarcinoma of the lung, with locally advanced or metastatic disease and not amenable to curative surgery or radiotherapy (stage IIIB, IIIC or IV disease based on the eighth edition of the American Joint Committee on Cancer (AJCC) TNM classification). Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
3. Patients must be treatment-naive for locally advanced or metastatic NSCLC systemic antitumor therapy. Prior adjuvant and neo-adjuvant therapy (except for EGFR-TKIs) is permitted if have been completed at least 6 months prior to initiation of disease progression.
4. Tissue or blood samples are confirmed by the central laboratory or research center as rare EGFR mutations, including exon 18 G719X, S768I in exon 20 and at least one of the L861Q mutations in exon 21;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Predicted survival ≥ 3 months.
7. At least 1 measurable tumor lesion without radiotherapy as per RECIST v1.1.
8. Agree to use effective contraception during the study period and for at least 3 months after completion of the study treatment.
9. Provision of informed consent prior to any study procedure.

Exclusion Criteria:

1. Combined with other malignancy(except for clinically cured in situ cervix carcinoma, basal cell or squamous epithelial skin cancer,thyroid papillary carcinoma).
2. Prior treatment with any EGFR-TKIs.
3. Prior treatment with any systemic antitumor therapy for locally advanced or metastatic NSCLC.
4. Previous traditional chinese medicine with an antitumor indication within 2 weeks before the first dose of study drug.
5. Previous major surgery within 4 weeks before the first dose of study drug,or planing to have major surgery during study.
6. Symptoms or signs worsened within 2 weeks before the first dose of study drug.
7. Any unresolved toxicities from prior treatment greater than NCI CTCAE v4.03 grade 2 or higher.
8. Spinal cord compression,symptomatic or unstable central nervous system (CNS) metastases that require the use of steroids .Patients who have a stable CNS status for at least 4 weeks before treatment will be allowed to join the study.
9. Any clinical evidence of serious or uncontrolled systemic disease,including uncontrolled hypertension after drug treatment,active bleeding diatheses, previous or present thrombus,uncontrolled cardiovascular and cerebrovascular diseases.
10. Active infection including hepatitis B,hepatitis C,syphilis and human immunodeficiency virus (HIV).
11. Mean resting corrected QT interval (QTcF) ≥450 msec,obtained from 3 ECGs or any clinically important abnormalities in rhythm,conduction, morphology of resting ECG or left ventricular ejection fraction (LVEF) ≤ 50%,etc.
12. Previous history of interstitial lung disease(ILD),drug-induced interstitial lung disease,history of radiation-induced pneumonia requiring hormone therapy,or clinical evidence of active interstitial lung disease.
13. Any instance that affects the patient's ability to swallow drug or oral malabsorption.
14. Occur any laboratory indicator abnormalities as follow：

    * absolute neutrophil count(ANC)<1,500/mcL
    * platelets<100,000/mcL
    * hemoglobin<9.0 g/dL
    * AST/ALT>2.5 times the upper limit of normal (ULN)or >5 times the ULN in the presence of liver metastases
    * total bilirubin(TBIL)>1.5 times the ULN if no liver metastases or > 3 times the ULN in the presence of liver metastases
    * serum creatinine(SCr) >1.5 times the ULN or creatinine clearance ≥50 mL/min.
15. Patients with a known allergy or delayed hypersensitivity reaction to the any component of study drugs or their excipients.
16. Within 1 week before the first dose of study drug currently receiving or need concomitant medications known to be potent inhibitors or inducers of CYP3A, CYP2D6,CYPC8 and CYP2C19,sensitive substrate of CYP3A and CYP2C9.
17. Within 1 week before the first dose of study drug ongoing use of warfarin.
18. Previous therapeutic clinical trial within 4 weeks before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | 24 months
  ORR, per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival（PFS） | 12 months
  PFS, defined as time from study drug administration to progression or death due to any cause.
Disease control rate（DCR） | 12 months
  DCR, defined as proportion of complete response, partial response, and disease stabilization to the proportion of patients with evalueable tumors.
Overall survival （OS） | 24 months
  OS, defined as the time from study drug administration until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes